CLINICAL TRIAL: NCT06330259
Title: Ist Die Konzentration Des Anti-Müllerschen Hormons (AMH) abhängig Vom Menstruationszyklus?
Brief Title: Does the AMH Concentration Depend on the Menstrual Cycle?
Acronym: AMH
Status: Completed | Type: Observational
Sponsor: University of Basel (Other)
Collaborators: Roche Diagnostics GmbH (Industry)
Responsible Party: Principal Investigator, Christian De Geyter, Prof., University of Basel
Other Study IDs: new AMH assay
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Reproductive Sterility
Keywords: natural menstrual cycle; AMH; 3D ultrasound
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: 25 younger women, aged 18 to 25 y.
  Interventions: Diagnostic Test: menstrual cycle monitoring
- Group B: 25 less young women, aged 26 to 39 y.
  Interventions: Diagnostic Test: menstrual cycle monitoring

INTERVENTIONS:
Diagnostic Test: menstrual cycle monitoring — frequent serum sampling and 3D ultrasound

SUMMARY:
During two none subsequent natural menstrual cycles healthy female participants will be subjected every second day to blood sampling and 3D-ultrasound examinations. Together with four other key hormones the concentration of AMH (anti-Muellerian Hormone) will be measured in the serum.

DETAILED DESCRIPTION:
During two none subsequent natural menstrual cycles healthy female participants will be subjected every second day to blood sampling and 3D-ultrasound examinations. Together with four other key hormones the concentration of AMH will be measured in the serum. Half of the serum samples will immediately be subjected to hormone analysis whereas the other half will be stored frozen at -80 °C. After conclusion of the study the frozen samples will be subjected to re-measurment again a reference laboratory. The aim is to study the stability of the AMH Elecsys Assay under both conditions. The participants will be health women aged between 18 and 40 years. They will be grouped into a younger and an older group. They will be observed during one menstrual cycle, then they will remain unobserved during a second menstrual cycle, and then again they will be observed during a third menstrual cycle.

ELIGIBILITY:
Inclusion Criteria:

* regular menstrual cycles, between 24 and 32 d.
* body mass index between 24 and 32 kg/m2
* no HIV, no Hepatitis B and C
* no smoking

Exclusion Criteria:

* intake of reproductive hormones, including birth control pill
* pregnancy or breastfeeding
* infertility
* polycystic ovary syndrome

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only women are recruited.
Study Population: healthy female women with regular menstrual cycles.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
AMH Elecsys Assay | 3 months
  The anti-Muellerian Hormone (AMH) is a heterodimer. As such, it is unstable. The newly developed assay is considered to account for this inherent instability of the hormone and is thought to produce more consistent results.

SECONDARY OUTCOMES:
Effect of handling of the serum on measured AMH concentrations | 3 months
  Handling of the serum samples may impact measured levels. The serum levels will be measured as part of daily routine both on the day of the sampling and in frozen samples (in batches, under maximal care conditions) the stability of observed serum values during the menstrual cycle
3D ultrasound of both ovaries | 3 months
  Fluctuations in the number of antral follicles during the menstrual cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Christian De Geyter, MD, Principal Investigator — University of Basel
Locations (1):
- Christian De Geyter, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No